CLINICAL TRIAL: NCT00116766
Title: Field Evaluation of Malaria Vector Control Using Traditional Plant-based Anti-mosquito Measures in Yunnan Province, P.R. China
Brief Title: Field Evaluation of Plant-based Mosquito Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Yunnan Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DIF28
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2007-02

CONDITIONS: Malaria; Arbovirus Infections
Keywords: mosquitoes; malaria; vector control; plant-based
MeSH Terms: conditions — Malaria; Arbovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: anti-mosquito plant use

SUMMARY:
Isolated minority communities in China use traditional plant-based methods of mosquito control. This study is evaluating 4 plants used in this way by monitoring mosquitoes entering houses on nights when the plants are being used in this way. A blind, placebo controlled study design will monitor plant use and record mosquito species / numbers caught in CDC light traps indoors over 3 months.

DETAILED DESCRIPTION:
Introduction

One of the greatest challenges to those planning vector control programmes in developing Countries is the provision of cover to those populations in remote or isolated areas. Commonly, it is these communities which bear the greatest burden of disease due to location and inaccessibility to local health care. Yunnan Province is a good example of such problems. The border region with Laos, Myanmar and Vietnam contributes a high proportion of all malaria cases in the whole of China, yet few if any disease control initiatives cover the rural minority peoples and migrant workers who inhabit the region. Comprehensive ethnobotanical surveys in the area have shown many of the 25 minority peoples living in isolated communities already use traditional herbal forms of mosquito control utilising several of the abundant species in the particularly diverse local environment. Having identified a number of potentially useful plant species being used, in terms of their availability, sustainability, low cost (free) and known chemical constituents, the investigators and the local Chinese malaria control officials consider a phase II evaluation of the most promising candidates is justified. In particular, 4 widely used plants are traditionally used as fumigants to reduce / prevent mosquitoes entering houses, either by burning dried or fresh material on the indoor cooking fires each evening, or by spraying tinctures around entry sites like eaves & windows. Due to the method of use, it would be very difficult to simulate this in the laboratory, so a simple means of field evaluation has been chosen.

Materials

The ethnobotanical survey revealed the following plant species as candidates for further study; Artemesia argyi, Eucalyptus robusta, Eupatorium odoratum, Cinnamomum glanduliferum

Each of these plant species occurs naturally in abundance in the region and collection will have no significant environmental impact. Moderate amounts (approx 1 Kg) sufficient for each study will be collected locally in each field site prior to (if used dried) or at the start of each experiment (fresh).

Methods

Plants will be evaluated under natural user conditions in a randomised and controlled manner in villages in Xishuangbanna Region, Yunnan, PR China. Village- based studies of several other mosquito control methods have already been successfully undertaken in this region by the LSHTM and YIPD team. Villages belonging to one of the ethnic groups using each traditional method will be selected according to agreement between local health workers from YIPD and the village elders, availability of plant species, and preliminary survey of vector species collected indoors with CDC traps. A different village will be selected for each plant being evaluated. After collecting background entomological data, 6 houses matched for baseline parameters (such as occupancy level, location, construction & animal proximity) and being evenly spaced among others in the village (to reduce diversion effects) will be enrolled into the study. On any one night, 2 will be allocated treatment (use of plant), 2 will be allocated hay (used for cattle bedding) as a negative control, and 2 will be left unused (to reduce any residual effects). In each case the treatment or control group will be instructed to place pre-prepared batches of plant material (weighed fresh or dry depending upon type) onto their cooking fire in the traditional manner in the early evening. Commercial CDC traps (BioQuip Inc., USA) will be used in / beside the sleeping areas of each house from 1 hour before sunset to early morning. Catches will be identified by local vector experts each day to record species and number. House treatment will be rotated each night using latin square principles to achieve a minimum of 12 replicates of each treatment in every house (36 nights duration, 216 trap/nights), and will take place during the rainy (malaria) season (July - Nov 2005) when both plants and vector levels are highest.

In the case of C. glanduliferum, the plant extract (or hay extract) will be sprayed at a predetermined rate onto eaves & doors / windows in the traditional manner following the same principles. Efficacy will be determined by comparing mosquito species / numbers caught in control & treatment houses using appropriate statistical analysis & ANOVA methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Existing use of traditional plant-based methods of mosquito control

Exclusion Criteria:

* Known allergy to plants in use
* Respiratory illness
* Infants under 6 years in house

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2005-07; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Reduction in vector mosquitoes entering houses | per night over 45 nights

SECONDARY OUTCOMES:
Reduced human biting by mosquitoes | per night over 45 nights

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Hill, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Hong Ning Zhou, MSc, Principal Investigator — Yunnan Institute of Parasitic Diseases